CLINICAL TRIAL: NCT05206929
Title: A Randomized Trial of Standard of Care Sternal Precautions VS Self Managed Care
Brief Title: Prescribed Sternal Precautions vs. Self-Guided Restrictive Care (PEEERC)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of current personnel availability. Plan to re-evaluate the study protocol and potentially reconsider study alterations in the future.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB20-1339
Record Dates: First submitted 2022-01-12; First posted 2022-01-25 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Surgery; Heart Diseases; Heart Failure; Cardiac Valve Disease
MeSH Terms: conditions — Heart Diseases; Heart Failure; Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Arm 1 will receive instruction to use pain and discomfort as the safe limits for their upper limb use during daily activities at post operative discharge.
  Interventions: Other: Self Managed Care
- Arm 2 (Active Comparator): Arm 2 will receive the standard sternal precautions at time of post operative discharge.
  Interventions: Other: Self Managed Care

INTERVENTIONS:
Other: Self Managed Care — Self Managed Care

SUMMARY:
Our study aims to compare postoperative outcomes, postoperative pain and postoperative quality of lives in patients who receive the standard sternal precautions to those in patients who received self-managed sternal precautions following sternotomy for cardiac surgeries. The purpose of the study is to see if self-managed sternal precautions following sternotomy for cardiac surgeries lead to better quality of lives while maintaining same postoperative pain and rate of postoperative adverse events than standard sternal precautions. Postoperative pain and postoperative quality of lives will be assessed by phone call surveys. Postoperative outcomes will be measured by following the patients for up to a year using electronic medical record.

DETAILED DESCRIPTION:
Patients who are recruited in this study will be randomized (1:1) into one of two groups/arms. The ?rst arm (Arm 1) will receive instruction to use pain and discomfort as the safe limits for their upper limb use during daily activities at post operative discharge. The second arm (Arm 2) will receive the standard sternal precautions at time of post operative discharge. Standard sternal precautions in study arm (2) include:

Don't reach both arms overhead Don't reach both arms out to the side Don't reach behind your back Don't lift more than 5 to 8 pounds Don't push with your arms Don't pull with your arms Don't drive

Each arm will receive weekly phone calls for 8 weeks. Information including pain, quality of life, and adherence to the sternal precaution protocol will be collected. Please refer to supporting documents (Pain Scale, Quality of Life Questionnaire, and Sternal Precaution Checklist) for the specific questions that will be asked at the patients. We will also investigate any adverse events related to the medical care.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a sternotomy, English speaking, 18-70 years old, able to ambulate independently

Exclusion Criteria:

* Sternotomy due to VAD implantation or cardiac transplantation, discharge over 1.5 weeks after surgery, prior sternotomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Sternal Precaution Checklist | Patient will be called weekly for 8 weeks by a medical professional.
  Assessing patients' adherence to protocol

SECONDARY OUTCOMES:
Sternal Precautions- Quality of Life Questions | Patient will be called weekly for 8 weeks by a medical professional.
  Assessing patients' postoperative quality of life
Sternal Precaution Pain Scale | Patient will be called weekly for 8 weeks by a medical professional.
  Assessing patients' postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: Valluvan Jeevanandam, MD, Principal Investigator — Professor of Surgery
Locations (1):
- The University of Chicago, Chicago, Illinois, United States